CLINICAL TRIAL: NCT07034586
Title: A Prospective Analysis of Adventitial Pathology in Patients Undergoing Coronary Bypass With Borderline Ascending Aortic Dilatation
Brief Title: Prospective Evaluation of Adventitial Histopathology in Borderline Ascending Aortic Dilatatio
Status: Active, not recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SUKAEK-2023 1/19
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ascending Aortic Aneurysm; Aortic Adventitial Pathology; Coronary Artery Bypass Grafting (CABG); Borderline Aortic Dilatation
Keywords: Aortic Dissection Risk Prediction; Borderline Aortic Dilatation; Ascending Aortic Aneurysm; Coronary Artery Bypass Grafting (CABG)
MeSH Terms: conditions — Aneurysm, Ascending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Aort Dilated Group: Patients undergoing elective coronary artery bypass grafting (CABG) with an ascending aortic diameter between 4.0 cm and 5.0 cm. These patients do not have known genetic aortopathy and are undergoing their first cardiac surgery. Aortic tissue samples are collected during surgery from the punch biopsy site used for proximal anastomosis.
- Observational Control Group: Patients undergoing elective CABG with an ascending aortic diameter less than 4.0 cm. These patients also do not have known aortopathies and are undergoing their first cardiac surgery. Punch biopsy material is similarly collected for histopathological evaluation.

SUMMARY:
This prospective study investigates microscopic changes in the outer layer (adventitia) of the ascending aorta in patients undergoing coronary artery bypass grafting (CABG) surgery. The study includes two groups of patients: (1) those with borderline ascending aortic dilatation (4.0-5.0 cm), and (2) a control group with normal aortic diameter (<4.0 cm), all undergoing the same surgical procedure. During CABG, a small circular punch is routinely made in the ascending aorta for the proximal saphenous vein graft anastomosis. The tissue removed from this punch site is collected and used for histopathological and immunohistochemical analysis. The study aims to determine whether adventitial changes correlate with aortic size and whether these changes can help identify patients at risk for future aortic dissection or rupture. The findings may guide surgical decision-making in patients with borderline aortic enlargement.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 20 and 70 years
2. Patients scheduled for elective open-heart coronary artery bypass grafting (CABG)
3. Patients undergoing their first cardiac surgery
4. Metabolically stable patients
5. Aortic diameter:

   1. Observational aortic dilatation group: between 4.0 cm and 5.0 cm
   2. Control group: less than 4.0 cm
6. Written informed consent obtained from the patient

Exclusion Criteria:

1. History of previous cardiac surgery
2. History of aortic dissection or rupture
3. Known genetic syndromes (e.g., Marfan, Loeys-Dietz, Ehlers-Danlos)
4. Known systemic vasculitis
5. Presence of acute infection or systemic inflammatory disease
6. Inadequate biopsy material for pathological analysis
7. Patients not undergoing any aortic intervention during surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 20 to 70 years undergoing elective coronary artery bypass grafting (CABG) surgery at a tertiary cardiovascular surgery center. Participants are divided into two groups based on preoperative ascending aortic diameter measured by imaging:
  Study Group: Patients with borderline ascending aortic dilatation (diameter between 4.0 cm and 5.0 cm) Control Group: Patients with normal ascending aortic diameter (<4.0 cm) All participants are undergoing their first cardiac surgery, are metabolically stable, and do not have a known history of aortic dissection, connective tissue disease, or systemic vasculitis.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Association Between Histopathological Findings and Aortic Diameter | Postoperative period (within 1 month)
  Comparison of adventitial tissue samples between patients with borderline ascending aortic dilatation (4.0-5.0 cm) and those with normal-sized aortas (<4.0 cm). Pathological evaluation includes staining for Carbonic Anhydrase IX (CA9), Smooth Muscle Actin (SMA), D2-40, Verhoeff-Van Gieson elastin, and Prussian blue. The presence of fibrosis, inflammation, neovascularization, and hypoxia-related markers will be recorded. Analysis of the correlation between the degree of histopathological changes and the measured ascending aortic diameter. Metrics include inflammatory cell infiltration, vasa vasorum density, and adventitial fibrosis severity.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Ereren, Study Chair — Samsun University Faculty of medicine
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided